CLINICAL TRIAL: NCT04870307
Title: Community-engaged Approaches to Testing in Community and Healthcare Settings for Underserved Populations
Acronym: CATCH-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12582; U54GM104938-08S1 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-05-03 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Covid19
Keywords: COVID-19; RADx-UP; Health Services Research; Implementation Science; Evidence-based practice; Social determinants of health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Dissemination and Implementation Research (D&I): Involves assisting primary care practices to address SARS-CoV-2 testing using evidence-based practices as well as increased testing in mobile-based community settings. The D&I model also involves Practice Assessment, Academic Detailing, Practice Facilitation, Health Information Technology Support, Performance Feedback and Benchmarking, and a Virtual Learning Community.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Care Practices (Other): A practice-based implementation study was conducted with 35 practices, with baseline data collection, and overlapping with interim measurements of care quality and process outcomes, followed by a final data collection at the end of the intervention. Patients were not direct subjects in this part of the study. The intervention targeted practices and practice members.
  Interventions: Other: Dissemination and Implementation Research

INTERVENTIONS:
Other: Dissemination and Implementation Research — Dissemination and Implementation research involves assisting primary care practices to address SARS-CoV-2 testing using evidence-based practices as well as increased testing in mobile-based community settings. The D&I model also involves Practice Assessment, Academic Detailing, Practice Facilitation, Health Information Technology Support, Performance Feedback and Benchmarking, and a Virtual Learning Community.

SUMMARY:
The pandemic caused by the novel coronavirus, Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), has resulted in substantial global morbidity and mortality including in Oklahoma and caused unprecedented interruptions in nearly all aspects of our lives. The population of the state of Oklahoma is at particular risk to SARS-CoV-2 due to its large rural population, strained healthcare system, and poor overall health. The Community-Engaged Approaches to Testing in Community and Healthcare Settings for Underserved Populations (CATCH-UP) program will involve both practice-based and community-based approaches to maximize the reach of the Rapid Acceleration of Diagnostics - Underserved Populations (RADx-UP) consortium, broaden the potential perspectives that could be captured, and compare the effectiveness of strategies. The interventions will be pragmatic to allow CATCH-UP to respond to changing attitudes, barriers, and environments as the pandemic progresses as well as expected technology developments to produce more effective viral testing that can provide rapid results to patients. The investigators will assist 50 small primary care practices to implement guidelines-based testing and patient education about Coronavirus Disease 2019 (COVID-19) and risk mitigation strategies. The project's community-based approach is designed to rapidly respond to community testing needs by deploying mobile testing sites that will provide operational support to increase the efficiency and the existing capacity for state-wide testing by Oklahoma's public health authorities. Together, the investigators estimate that the CATCH-UP program will result in at least 105,000 SARS-CoV-2 tests performed during the first year of implementation. A comprehensive, ongoing evaluation will be performed to analyze patient and provider attitudes, barriers and facilitators of viral testing, identified health disparities caused by COVID-19, effectiveness of the intervention in both settings, and to allow robust collaboration with other RADx-UP consortium sites.

DETAILED DESCRIPTION:
The broad RADx-UP initiative aims to understand the factors associated with COVID-19 morbidity and mortality disparities and to lay the foundation to reduce disparities for underserved and vulnerable populations disproportionately affected by the pandemic through efforts to increase access and effectiveness of diagnostic methods. The approach used in this project will leverage the investigators' experiences in designing and implementing evidence-based interventions in primary care settings, partnerships with Native American and Latino communities, investments in the development of community- driven and responsive organizations developed primarily in rural counties, and the capacity and needs of Oklahoma's government testing and contact tracing infrastructure to develop, test, and evaluate a culturally- responsive SARS-CoV-2 testing intervention, collection of additional data on COVID-19 related health disparities, and identification of additional attitudes, facilitators, and barriers to testing and eventual vaccination.

The investigators have designed an approach that not only allows for collecting essential information about community, provider, and patient-relevant impediments to viral testing but also meeting the critical need to increase testing in testing deserts in Oklahoma as rapidly as possible. The investigators believe that a singular focus on one testing strategy will be ineffective in truly understanding the barriers to testing. No one strategy would be effective in reaching all of the population, due to issues such as lack of access to a primary care provider, lack of insurance, transportation, available time, or individual/community perceptions on testing itself (e.g., safety, necessity, availability, trust). Thus, the investigators have chosen to develop the Community-engaged Approaches to Testing in Community and Healthcare settings for Underserved Populations (CATCH-UP) program with practice-based and community-based approaches to maximize the reach of the RADx-UP consortium, broaden the potential perspectives that could be captured, and compare the effectiveness of strategies. Rather than developing an inflexible practice-based intervention a priori, the investigators believe that the ever-changing barriers, attitudes and conditions in the pandemic, as well as the development and deployment of more effective diagnostic technologies over the next few months, necessitate a pragmatic approach in which increased testing is initiated quickly while simultaneously collaborating with stakeholders and collecting participant survey data in real-time, which will allow the intervention to evolve to changing needs, and provide rapid-cycle evaluation of effectiveness of these activities to provide timely feedback to the partners and other RADx-UP initiatives.

The specific aims of the CATCH-UP Project are as follows:

1. Provide technical support to a minimum of 50 Oklahoma primary care practices to implement a person-centered approach to SARS-CoV-2 testing based on best available evidence and current guidelines. The implementation approach will include 1) development of implementation support resources for COVID-19 testing and risk mitigation strategies to meet the needs of vulnerable populations through continuous adaption to changing guidelines, testing protocols and availability, and information learned from the project's provider network and the broader RADx-UP community, 2) support practices to integrate tailored, guideline- based SARS-CoV-2 testing protocols and resources into the workflows through proven methodologies of academic detailing from peer-physician experts, practice change facilitation through quality improvement implementation professionals, and health information technology support. Based on the average number of providers and daily caseload in rural Oklahoma practices the investigators estimate this will result in approximately 60,000 viral tests performed in the first year.
2. Rapidly respond to community testing needs by deploying mobile testing units in community settings that will provide operational support to increase the efficiency and the existing capacity for statewide testing by Oklahoma's public health authorities. The model used by the Chickasaw Nation in deploying a high-efficiency community testing system will be combined with ongoing observation and analysis to identify facilitators and barriers to implementing community testing sites to accelerate convergence on effective and replicable methods to increase access and acceptance of testing. The investigators will adapt to ongoing disease outbreaks and community needs, but anticipate that this aim will result in more than 250 testing events at sites throughout the state and 45,000 viral tests performed in the first year.
3. Conduct a comprehensive evaluation of the impact of the CATCH-UP program, collaborate closely with other RADx-UP projects in sharing data and adapting processes, and continuously communicate with our community partners to assess effectiveness and disseminate research findings. This evaluation will include measurement and dissemination of data related to 1) Provider-level Outcomes that include knowledge and attitudes of disease prevalence, clinical characteristics including typical and atypical symptoms and disease severity, testing importance and strategies, vaccination, importance and use of personal protective equipment, availability of testing and delays in return of results, and provider observations of patient attitudes and other reported barriers, 2) Care Process Outcomes such as testing, test positivity, and test refusal rates, influenza, pneumococcal, and zoster vaccination rates, 3) Community-level Outcomes that include the number of tests conducted by mobile testing units and the resulting test positivity rate, 4) Patient-level Outcomes such as knowledge and attitudes of disease prevalence, disease characteristics including severity and acute and chronic symptoms, risk perspective and preferences, importance and use of personal protective equipment, patient acceptance of various testing options, and facilitators and barriers to participating in testing and future vaccination programs, 5) Patient Factors such as demographics, social determinants of health, and clinical characteristics that may be associated with COVID-19 morbidity and mortality disparities or reach of each testing modality, and 6) Qualitative Outcomes including perceptions of facilitators and barriers to testing and the utility, effectiveness, and generalizability of the program, explored through key informant interviews, exit interviews, and in-depth program implementation process observations.

ELIGIBILITY:
Inclusion Criteria:

* Practices:

  1. Primary care practices located in Oklahoma.
  2. Priority to practices serving a majority of patients that are underserved or vulnerable populations (rural, minority, elderly).
  3. Practices routinely using a certified electronic health record (EHR) will be eligible to participate, as practices that are still using paper records are either planning to close due to clinician retirement or will likely be implementing an EHR during the project, which would compromise their ability to participate.
  4. Practice-wide participation will be encouraged, but participation of all members within a practice (both clinicians and staff members) will not be required. The minimum acceptable level of participation will be one clinician and nurse/medical assistant dyad plus anyone else who would have to be involved to make changes in the processes of care (e.g. clinic manager) for that unit of care.
  5. Clinicians and staff members 18 years of age and older at the time of enrollment (consent).
* Patients survey participants:

  1. Patients (or caregivers of patients) who are seen in eligible practices or community testing sites and received a recommendation for the patient to receive a SARS-CoV-2 diagnostic test.
  2. Patients (or their caregivers) who are 18 or older

Exclusion Criteria:

* Practices:

  1. Practices that are uninterested in reducing missed opportunities for guidelines-based testing for SARS-CoV-2
  2. Solo practices with a clinician planning to retire within 12 months of enrollment will not be eligible for participation.
  3. Practices likely to experience ownership change in the next 12 months will not be eligible for participation.
* Patient survey participants:

  1. Patients unable to complete the consent process or survey instruments in English or Spanish.
  2. Patients or caregivers of patients who are under the age of 18.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A James, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma Clinical and Translational Science Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDC COVID-19 Response Team. Geographic Differences in COVID-19 Cases, Deaths, and Incidence - United States, February 12-April 7, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):465-471. doi: 10.15585/mmwr.mm6915e4. PMID 32298250
- [Background] Zhang CH, Schwartz GG. Spatial Disparities in Coronavirus Incidence and Mortality in the United States: An Ecological Analysis as of May 2020. J Rural Health. 2020 Jun;36(3):433-445. doi: 10.1111/jrh.12476. Epub 2020 Jun 16. PMID 32543763
- [Background] Shahid Z, Kalayanamitra R, McClafferty B, Kepko D, Ramgobin D, Patel R, Aggarwal CS, Vunnam R, Sahu N, Bhatt D, Jones K, Golamari R, Jain R. COVID-19 and Older Adults: What We Know. J Am Geriatr Soc. 2020 May;68(5):926-929. doi: 10.1111/jgs.16472. Epub 2020 Apr 20. PMID 32255507
- [Background] Iaccarino G, Grassi G, Borghi C, Ferri C, Salvetti M, Volpe M; SARS-RAS Investigators. Age and Multimorbidity Predict Death Among COVID-19 Patients: Results of the SARS-RAS Study of the Italian Society of Hypertension. Hypertension. 2020 Aug;76(2):366-372. doi: 10.1161/HYPERTENSIONAHA.120.15324. Epub 2020 Jun 22. PMID 32564693
- [Background] CDC COVID-19 Response Team. Preliminary Estimates of the Prevalence of Selected Underlying Health Conditions Among Patients with Coronavirus Disease 2019 - United States, February 12-March 28, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):382-386. doi: 10.15585/mmwr.mm6913e2. PMID 32240123
- [Background] Wang X, Fang X, Cai Z, Wu X, Gao X, Min J, Wang F. Comorbid Chronic Diseases and Acute Organ Injuries Are Strongly Correlated with Disease Severity and Mortality among COVID-19 Patients: A Systemic Review and Meta-Analysis. Research (Wash D C). 2020 Apr 19;2020:2402961. doi: 10.34133/2020/2402961. eCollection 2020. PMID 32377638
- [Background] Turner-Musa J, Ajayi O, Kemp L. Examining Social Determinants of Health, Stigma, and COVID-19 Disparities. Healthcare (Basel). 2020 Jun 12;8(2):168. doi: 10.3390/healthcare8020168. PMID 32545647
- [Background] Rollston R, Galea S. COVID-19 and the Social Determinants of Health. Am J Health Promot. 2020 Jul;34(6):687-689. doi: 10.1177/0890117120930536b. No abstract available. PMID 32551932
- [Background] Hawkins D. Differential occupational risk for COVID-19 and other infection exposure according to race and ethnicity. Am J Ind Med. 2020 Sep;63(9):817-820. doi: 10.1002/ajim.23145. Epub 2020 Jun 15. PMID 32539166
- [Background] Terry DL, Woo MJ. Burnout, job satisfaction, and work-family conflict among rural medical providers. Psychol Health Med. 2021 Feb;26(2):196-203. doi: 10.1080/13548506.2020.1750663. Epub 2020 Apr 13. PMID 32281405
- [Background] Kaufman BG, Whitaker R, Pink G, Holmes GM. Half of Rural Residents at High Risk of Serious Illness Due to COVID-19, Creating Stress on Rural Hospitals. J Rural Health. 2020 Sep;36(4):584-590. doi: 10.1111/jrh.12481. Epub 2020 Jun 30. PMID 32603030
- [Background] Davoodi NM, Healy M, Goldberg EM. Rural America's Hospitals are Not Prepared to Protect Older Adults From a Surge in COVID-19 Cases. Gerontol Geriatr Med. 2020 Jul 7;6:2333721420936168. doi: 10.1177/2333721420936168. eCollection 2020 Jan-Dec. PMID 32685610
- [Background] James CV, Moonesinghe R, Wilson-Frederick SM, Hall JE, Penman-Aguilar A, Bouye K. Racial/Ethnic Health Disparities Among Rural Adults - United States, 2012-2015. MMWR Surveill Summ. 2017 Nov 17;66(23):1-9. doi: 10.15585/mmwr.ss6623a1. PMID 29145359
- [Background] Henning-Smith C, Tuttle M, Kozhimannil KB. Unequal Distribution of COVID-19 Risk Among Rural Residents by Race and Ethnicity. J Rural Health. 2021 Jan;37(1):224-226. doi: 10.1111/jrh.12463. Epub 2020 Jun 25. No abstract available. PMID 32396220
- [Background] Bavel JJV, Baicker K, Boggio PS, Capraro V, Cichocka A, Cikara M, Crockett MJ, Crum AJ, Douglas KM, Druckman JN, Drury J, Dube O, Ellemers N, Finkel EJ, Fowler JH, Gelfand M, Han S, Haslam SA, Jetten J, Kitayama S, Mobbs D, Napper LE, Packer DJ, Pennycook G, Peters E, Petty RE, Rand DG, Reicher SD, Schnall S, Shariff A, Skitka LJ, Smith SS, Sunstein CR, Tabri N, Tucker JA, Linden SV, Lange PV, Weeden KA, Wohl MJA, Zaki J, Zion SR, Willer R. Using social and behavioural science to support COVID-19 pandemic response. Nat Hum Behav. 2020 May;4(5):460-471. doi: 10.1038/s41562-020-0884-z. Epub 2020 Apr 30. PMID 32355299
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Linton NM, Kobayashi T, Yang Y, Hayashi K, Akhmetzhanov AR, Jung SM, Yuan B, Kinoshita R, Nishiura H. Incubation Period and Other Epidemiological Characteristics of 2019 Novel Coronavirus Infections with Right Truncation: A Statistical Analysis of Publicly Available Case Data. J Clin Med. 2020 Feb 17;9(2):538. doi: 10.3390/jcm9020538. PMID 32079150
- [Background] Furukawa NW, Brooks JT, Sobel J. Evidence Supporting Transmission of Severe Acute Respiratory Syndrome Coronavirus 2 While Presymptomatic or Asymptomatic. Emerg Infect Dis. 2020 Jul;26(7):e201595. doi: 10.3201/eid2607.201595. Epub 2020 Jun 21. PMID 32364890
- [Background] Arons MM, Hatfield KM, Reddy SC, Kimball A, James A, Jacobs JR, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Dyal JW, Harney J, Chisty Z, Bell JM, Methner M, Paul P, Carlson CM, McLaughlin HP, Thornburg N, Tong S, Tamin A, Tao Y, Uehara A, Harcourt J, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Montgomery P, Stone ND, Clark TA, Honein MA, Duchin JS, Jernigan JA; Public Health-Seattle and King County and CDC COVID-19 Investigation Team. Presymptomatic SARS-CoV-2 Infections and Transmission in a Skilled Nursing Facility. N Engl J Med. 2020 May 28;382(22):2081-2090. doi: 10.1056/NEJMoa2008457. Epub 2020 Apr 24. PMID 32329971
- [Background] Tromberg BJ, Schwetz TA, Perez-Stable EJ, Hodes RJ, Woychik RP, Bright RA, Fleurence RL, Collins FS. Rapid Scaling Up of Covid-19 Diagnostic Testing in the United States - The NIH RADx Initiative. N Engl J Med. 2020 Sep 10;383(11):1071-1077. doi: 10.1056/NEJMsr2022263. Epub 2020 Jul 22. No abstract available. PMID 32706958
- [Background] Dwyer JW, Contreras D, Eschbach CL, Tiret H, Newkirk C, Carter E, Cronk L. Cooperative Extension as a Framework for Health Extension: The Michigan State University Model. Acad Med. 2017 Oct;92(10):1416-1420. doi: 10.1097/ACM.0000000000001640. PMID 28353501
- [Background] Grumbach K, Mold JW. A health care cooperative extension service: transforming primary care and community health. JAMA. 2009 Jun 24;301(24):2589-91. doi: 10.1001/jama.2009.923. No abstract available. PMID 19549977
- [Background] Kaufman A, Boren J, Koukel S, Ronquillo F, Davies C, Nkouaga C. Agriculture and Health Sectors Collaborate in Addressing Population Health. Ann Fam Med. 2017 Sep;15(5):475-480. doi: 10.1370/afm.2087. PMID 28893819
- [Background] Phillips RL Jr, Kaufman A, Mold JW, Grumbach K, Vetter-Smith M, Berry A, Burke BT. The primary care extension program: a catalyst for change. Ann Fam Med. 2013 Mar-Apr;11(2):173-8. doi: 10.1370/afm.1495. PMID 23508605
- [Background] Chou AF, Homco JB, Nagykaldi Z, Mold JW, Daniel Duffy F, Crawford S, Stoner JA. Disseminating, implementing, and evaluating patient-centered outcomes to improve cardiovascular care using a stepped-wedge design: healthy hearts for Oklahoma. BMC Health Serv Res. 2018 Jun 4;18(1):404. doi: 10.1186/s12913-018-3189-4. PMID 29866120
- [Background] Bodenheimer T, Ghorob A, Willard-Grace R, Grumbach K. The 10 building blocks of high-performing primary care. Ann Fam Med. 2014 Mar-Apr;12(2):166-71. doi: 10.1370/afm.1616. PMID 24615313
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Kenney C. Transforming Health Care. Virginia Mason Medical Center's Pursuit of the Perfect Patient Experience.: Productivity Press.; 2010
- [Background] Chao EC. Structured correlation in models for clustered data. Stat Med. 2006 Jul 30;25(14):2450-68. doi: 10.1002/sim.2368. PMID 16220520
- [Background] van Oest R. A new coefficient of interrater agreement: The challenge of highly unequal category proportions. Psychol Methods. 2019 Aug;24(4):439-451. doi: 10.1037/met0000183. Epub 2018 May 3. PMID 29723005
- [Background] Cohen DJ, Crabtree BF. Evaluative criteria for qualitative research in health care: controversies and recommendations. Ann Fam Med. 2008 Jul-Aug;6(4):331-9. doi: 10.1370/afm.818. PMID 18626033
- See also: Abrams EM, Szefler SJ. COVID-19 and the impact of social determinants of health. The Lancet Respiratory Medicine. 2020;8(7):659-61. doi: 10.1016/s2213-2600(20)30234-4. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7234789/
- See also: 2020 Rural Hospital Sustainability Index 2020 [cited 2020] — https://guidehouse.com/insights/healthcare/2020/rural-hospital-sustainability-index
- See also: United States Department of Agriculture ERS. State Fact Sheet: United States. — https://data.ers.usda.gov/reports.aspx?ID=17854
- See also: United States Department of Agriculture ERS. State Fact Sheets: Oklahoma — https://data.ers.usda.gov/reports.aspx?StateFIPS=40&StateName=Oklahoma&ID=17854
- See also: Oklahoma Primary Healthcare Improvement Cooperative (OPHIC). The Research to Practice to Research Exchange 2018 — https://rpr.lib.ok.us/library
- See also: Scoville R, Little K. Comparing Lean and Quality Improvement. IHI White Paper. Cambridge, MA: Institute for Healthcare Improvement; 2014 — https://www.ihi.org/resources/white-papers/comparing-lean-and-quality-improvement
- See also: Grayson K, R. R. Interrater Reliability. Journal of Consumer Psychology. 2001;10(1):71-3. doi: 10.1207/15327660151043998 — https://scholar.google.com/citations?view_op=view_citation&hl=en&user=wFNeuYwAAAAJ&citation_for_view=wFNeuYwAAAAJ:uWQEDVKXjbEC

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Practices
Groups:
- Primary Care Practices: A practice-based implementation study was conducted with 35 primary care practices, with baseline data collection, and overlapping interim measurements of care quality and process outcomes, followed by a final data collection at the end of the intervention.
  The practice-based approach involved assisting primary care practices to address SARS-CoV-2 testing using evidence-based practices. The intervention model included practice assessment, academic detailing, practice facilitation, health information technology support, performance feedback and benchmarking, and a virtual learning community.
  Practice members were surveyed to better understand barriers to SARS-CoV-2 testing. Patients were not direct subjects. The intervention targeted practices and practice members.
Period: Overall Study
Arm/Group | Primary Care Practices
Started | 323; 35 Practices
Completed | 149; 22 Practices
Not Completed | 174; 13 Practices

BASELINE CHARACTERISTICS:
Population: Participants are primary care practice members within the 35 participating practices (physicians, physician assistants, nurse practitioners, clinical staff, office managers, etc.)
Units Other Than Participants: Practices
Groups:
- Primary Care Practices: A practice-based implementation study was conducted with 35 practices, with baseline data collection, and overlapping with interim measurements of care quality and process outcomes, followed by a final data collection at the end of the intervention (including baseline measures plus semi-structured interviews. The practice based approach to increasing testing will be compared to a community-based approach using mobile-setting to increase testing. Additional, non-clinical trial components of this study include patient surveys to understand facilitators and barriers to SARS-CoV-2 testing and identification of legal/ethical, socioeconomic, and behavioral implications of increased testing. Patients are not direct subjects in this part of the study. Intervention will target practices and practice members.
  Dissemination and Implementation Research: Dissemination and Implementation research involves assisting primary care practices to address SARS-CoV-2 testing using evidence-based practices as well as increased testing in mobile-based community settings. The D&I model also involves Practice Assessment, Academic Detailing, Practice Facilitation, Health Information Technology Support, Performance Feedback and Benchmarking, and a Virtual Learning Community.
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 323
Number analyzed (Practices) | 35
Age, Categorical [Count of Participants; unit: Participants] — Population: Age information was only collected for 179 participants.
  Participants
    number analyzed (Participants) | 179
    <=18 years | 0
    Between 18 and 65 years | 168
    >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information for sex (female/male) was not collected for 128 participants.
  Participants
    number analyzed (Participants) | 195
    Female | 172
    Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 151
  More than one race | 23
  Unknown or Not Reported | 125
Region of Enrollment [Number; unit: participants]
  United States | 323

OUTCOME MEASURES:

1. Primary Outcome: Change in SARS-CoV-2 Testing Rate (Practices)
Description: Change in the proportion of patients eligible for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) testing based on screening that receive SARS-CoV-2 test. The proportion ranges between zero and one.
Time Frame: Baseline to 12 months
Population: The average proportion of patients receiving a SARS-CoV-2 test at the practice-level. Data were collected at the practice level only, no participant or patient level data were collected.
Measure: Mean (Standard Deviation); unit: proportion of patients (ranging 0-1)
Units Other Than Participants: Practices
Groups:
- Primary Care Practices: A practice-based implementation study was conducted with 35 practices, with baseline data collection, and overlapping with interim measurements, followed by a final data collection at the end of the intervention. Patients are not direct subjects in this part of the study. The intervention targeted practices and practice members.
Arm/Group | Primary Care Practices
Number analyzed (Participants) | NA
Number analyzed (Practices) | 22
proportion of patients (ranging 0-1)
  Baseline | 0.9928 (0.0348)
  12 months | 1 (0)

2. Primary Outcome: Change in SARS-CoV-2 Test Positivity Rate
Description: Change in the proportion of SARS-CoV-2 test results that are positive.
Time Frame: Baseline to 12 months
Population: The proportion of SARS-CoV-2 tests conducted at each participating practice that were positive were recorded at both baseline and at 12 months. These practice-level proportions were averaged. Data were collected at the practice level only, no participant or patient level data were collected.
Measure: Mean (Standard Deviation); unit: proportion of tests (ranging 0-1)
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | NA
Number analyzed (Practices) | 23
proportion of tests (ranging 0-1)
  Baseline | 0.0660 (0.0972)
  12 Months | 0.2545 (0.1862)

3. Primary Outcome: Barriers to SARS-CoV-2 Testing
Description: Number (and type) of barriers to SARS-CoV-2 testing reported by practice members based on what they experienced during practice encounters with patients during the study.
Time Frame: Baseline
Population: Primary care practice members reported barriers to SARS-CoV-2 testing on a Practice Member Survey. Practice members could report more than one barrier.
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 244
Number analyzed (Practices) | 35
participants
  Not feeling sick therefore not wanting to be tested | 134
  Testing not available | 41
  Fear of receiving nasopharyngeal testing | 119
  Transportation | 69
  Not being able to pay | 95
  Not knowing where to go for testing | 87
  Childcare | 67
  Not able to take time off work | 116

4. Primary Outcome: Barriers to SARS-CoV-2 Testing (Practices)
Description: as for outcome 3
Time Frame: Month 3
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 110
Number analyzed (Practices) | 28
participants
  Not feeling sick therefore not wanting to be tested | 62
  Testing not available | 3
  Fear of receiving nasopharyngeal testing | 58
  Transportation | 27
  Not being able to pay | 27
  Not knowing where to go for testing | 22
  Childcare | 19
  Not able to take time off work | 45
  Already had COVID-19 and don't think testing is needed | 58
  Don't see testing as important | 29

5. Primary Outcome: Barriers to SARS-CoV-2 Testing (Practices)
Description: as for outcome 3
Time Frame: Month 6
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 125
Number analyzed (Practices) | 26
participants
  Not feeling sick therefore not wanting to be tested | 59
  Testing not available | 5
  Fear of receiving nasopharyngeal testing | 45
  Transportation | 23
  Not being able to pay | 28
  Not knowing where to go for testing | 17
  Childcare | 25
  Not able to take time off work | 45
  Already had COVID-19 and don't think testing is needed | 63
  Don't see testing as important | 34

6. Primary Outcome: Barriers to SARS-CoV-2 Testing (Practices)
Description: as for outcome 3
Time Frame: Month 9
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 114
Number analyzed (Practices) | 25
participants
  Not feeling sick therefore not wanting to be tested | 60
  Testing not available | 7
  Fear of receiving nasopharyngeal testing | 45
  Transportation | 27
  Not being able to pay | 21
  Not knowing where to go for testing | 12
  Childcare | 27
  Not able to take time off work | 42
  Already had COVID-19 and don't think testing is needed | 68
  Don't see testing as important | 43

7. Primary Outcome: Barriers to SARS-CoV-2 Testing (Practices)
Description: as for outcome 3
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 111
Number analyzed (Practices) | 22
participants
  Not feeling sick therefore not wanting to be tested | 48
  Testing not available | 3
  Fear of receiving nasopharyngeal testing | 39
  Transportation | 24
  Not being able to pay | 16
  Not knowing where to go for testing | 9
  Childcare | 25
  Not able to take time off work | 48
  Already had COVID-19 and don't think testing is needed | 56
  Don't see testing as important | 39

8. Secondary Outcome: Change in Influenza Vaccination Rate (NQF #41)
Description: Change in the proportion of patients aged 6 months and older who received an influenza immunization or reported receipt of an influenza immunization. Influenza Vaccination Rate was defined in alignment with National Quality Forum (NQF) measure #41 and was recorded as a proportion ranging between zero and one.
Time Frame: Baseline to 12 months
Population: Proportion of patients receiving influenza vaccine at the practice-level at baseline versus at 12 months. Data were collected at the practice level only, no participant or patient level data were collected.
Measure: Mean (Standard Deviation); unit: proportion of patients (ranging 0-1)
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | NA
Number analyzed (Practices) | 7
proportion of patients (ranging 0-1)
  Baseline | 0.2376 (0.2051)
  12 Months | 0.1110 (0.1701)

9. Secondary Outcome: Change in Pneumococcal Vaccination Rate (NQF #127)
Description: Change in the proportion of patients 65 years of age or older who have ever received a pneumococcal vaccine. Pneumococcal Vaccination Rate was defined in alignment with National Quality Forum (NQF) measure #41 and was recorded as a proportion ranging between zero and one.
Time Frame: Baseline to 12 months
Population: Proportion of patients receiving pneumococcal vaccine at the practice-level at baseline versus at 12 months. Data were collected at the practice level only, no participant or patient level data were collected.
Measure: Mean (Standard Deviation); unit: proportion of patients (ranging 0-1)
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | NA
Number analyzed (Practices) | 7
proportion of patients (ranging 0-1)
  Baseline | 0.1240 (0.1749)
  12 Months | 0.1053 (0.1805)

10. Secondary Outcome: Change in Zoster Vaccination Rate
Description: Change in the proportion of patients aged 50 years and older who have had the Shingrix zoster (shingles) vaccination. Proportion ranges from zero to one.
Time Frame: Baseline to 12 months
Population: Data were not collected because collection of Zoster vaccination rates from primary care practices requires an electronic medical record query that was not available across participating practices.
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 0

11. Secondary Outcome: COVID-19 Referrals
Description: Practices that reported not administering the COVID-19 vaccine were asked "Where do you send your patients that require a COVID-19 vaccine?" on the Practice Member Survey.
Time Frame: Baseline
Population: The plan was to report where primary care practices reported referring patients to for the COVID-19 vaccine, but data were not collected for this time frame.
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 0

12. Secondary Outcome: COVID-19 Referrals
Description: as for outcome 11
Time Frame: Month 3
Population: as for outcome 11
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 0

13. Secondary Outcome: COVID-19 Referrals
Description: as for outcome 11
Time Frame: Month 6
Population: Primary care practice members reported where they refer patients to for the COVID-19 vaccine. Note, practice members could report more than one referral location.
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 68
Number analyzed (Practices) | 18
participants
  Local health department | 51
  Pharmacy | 50
  Other provider in health system | 10
  Other | 5

14. Secondary Outcome: COVID-19 Referrals
Description: as for outcome 11
Time Frame: Month 9
Population: as for outcome 13
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 68
Number analyzed (Practices) | 17
participants
  Local health department | 56
  Pharmacy | 56
  Other provider in health system | 7
  Other | 2

15. Secondary Outcome: COVID-19 Referrals
Description: as for outcome 11
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: participants
Units Other Than Participants: Practices
Arm/Group | Primary Care Practices
Number analyzed (Participants) | 56
Number analyzed (Practices) | 17
participants
  Local health department | 46
  Pharmacy | 36
  Other provider in health system | 5
  Other | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 29 months
Description: All-cause mortality was tracked for enrolled participants starting at participant enrollment and throughout their participation in the study.
Groups:
- Primary Care Practices: A practice-based implementation study was conducted with 35 practices, with baseline data collection, and overlapping with interim measurements of care quality and process outcomes, followed by a final data collection at the end of the intervention including baseline measures plus semi-structured interviews. The practice based approach to increasing testing will be compared to a community-based approach using mobile-setting to increase testing. Additional, non-clinical trial components of this study include patient surveys to understand facilitators and barriers to SARS-CoV-2 testing and identification of legal/ethical, socioeconomic, and behavioral implications of increased testing. Patients are not direct subjects in this part of the study. Intervention will target practices and practice members.
  Dissemination and Implementation Research: Dissemination and Implementation research involves assisting primary care practices to address SARS-CoV-2 testing using evidence-based practices as well as increased testing in mobile-based community settings. The D&I model also involves Practice Assessment, Academic Detailing, Practice Facilitation, Health Information Technology Support, Performance Feedback and Benchmarking, and a Virtual Learning Community.
Arm/Group | Primary Care Practices
All-Cause Mortality (participants affected / at risk) | 2/323
Serious Adverse Events (participants affected / at risk) | 0/323
Other Adverse Events (participants affected / at risk) | 0/323

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04870307/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04870307/SAP_001.pdf
  • Informed Consent Form (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04870307/ICF_002.pdf